CLINICAL TRIAL: NCT06222346
Title: Online Peer Support in Long-term Conditions: a Feasibility Randomised Controlled Trial
Brief Title: Online Peer Support in Long-term Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: BitJam (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 328175
Record Dates: First submitted 2023-06-20; First posted 2024-01-24 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-07

CONDITIONS: Long-term Physical Health Conditions; Subthreshold Depression
Keywords: online; peer support; psychoeducation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CommonGround Platform (Experimental): Online Peer Support and Psychoeducational Platform
  Interventions: Behavioral: CommonGround
- Control (Active Comparator): National Health Service (NHS) "Mental Health" webpage(s)
  Interventions: Behavioral: NHS Mental Health

INTERVENTIONS:
Behavioral: CommonGround — Through collaboration with people living with LTCs, clinicians, academics, and web design experts, we have co-designed an online peer support and psychoeducation platform to help people with physical health conditions connect, support others, share experiences, and receive evidence-based information and advice on self-management. The web-based platform offers users access to peer support forums with embedded psychoeducation content.
  The following components are key features of the platform:
  * A discussion forum
  * A private "My Garden" page that stores posts from other users and psychoeducation content that the user has decided to 'save'.
  * A "resources" page giving access to evidence-based psychoeducation material on the mind-body link
  * A 'Crisis and Further Support' page, where users can find further organisations and sources of support, particularly for crisis situations. The peer support platform does not offer one-to-one or crisis support.
  Arms: CommonGround Platform
Behavioral: NHS Mental Health — Participants in the control arm will be directed towards the "Mental Health" webpage(s), an online resources page provided by the NHS. These resources are not specifically targeted at people living with LTCs. They include information sheets and mental health support on topics such as advice for life situations and events. Additionally, it hosts a "self-help" section that includes guides, tools, and activities to support mental health, but does not include any interactive or peer support elements.
  Arms: Control

SUMMARY:
Over 15 million people in England live with a long-term physical health condition. Low mood, loneliness and worry related to chronic illness are very common. In partnership with people with long-term conditions we have co-designed an online peer support platform to help people with health problems connect, support others, share experiences, and receive evidence-based information and advice on self-management.

This study explores if the platform is feasible to implement and acceptable for people with long-term conditions experiencing mild depressive symptoms. Those allocated to the intervention arm will be invited to try out an online peer support platform with psychoeducational resources named "CommonGround". Those in the control arm will be guided to use the National Health Service NHS "Mental Health" webpages.

DETAILED DESCRIPTION:
Approximately 20% of people with a long-term conditions (LTC) experience subthreshold depression (SUBD), which is also a key risk factor for developing more significant depression. There is currently no targeted psychological support for people with LTC also experiencing SUBD. This work offers a potentially novel way of addressing this gap through the delivery of an online peer support and psychoeducation platform. This project builds on previously funded work, which has enabled the co-production of a platform curated through cross-collaborations of people with LTC, clinicians, academics, and web design experts.

Study Design:

This is a mixed method, two-arm, parallel group, unblinded randomised controlled feasibility trial, with nested qualitative interviews evaluating participant experiences.

Population, Study Setting and Recruitment:

People living with long-term conditions who are experiencing subthreshold depression will take part in the randomised controlled trial. All participants will be recruited in the United Kingdom by King's College London (KCL). Both treatment arms will be delivered online. Participants will be randomly allocated to receive either the intervention (peer support and psychoeducation platform) or a control condition.

Recruitment:

Five routes will be used for recruitment. The feasibility of recruiting through each of these listed recruitment avenues will be assessed.

Routes 1: We will recruit participants with LTCs and SUBD from outpatient clinics at King's College Hospital NHS Foundation Trust and Guy's and St Thomas's NHS Foundation Trust that have used the IMPARTS platform. Clinicians in IMPARTS clinics will share information sheets with potentially suitable patients, and flyers will be displayed in waiting rooms, to invite interested participants to contact the research team directly.

Route 2: Other consent to contact patient databases (e.g., The BioResource database; IAPT Lambeth Talking Therapies). The research team or gatekeepers from these organisations will contact individuals to share the information sheet and eligibility screening with those who have consented to contact.

Route 3: Outpatient clinics at King's College Hospital NHS Foundation Trust and Guy's and St Thomas's NHS Foundation Trust where IMPARTS has not been implemented will be approached to facilitate recruitment. Other primary or secondary care settings may also be approached (e.g., GP practices, other NHS Trusts with specialised clinics for long-term conditions). Clinic staff will offer patients information sheets and display flyers in waiting rooms, inviting interested participants to contact the research team directly to register their interest or access the online participant information sheet.

Route 4: Public advertisements will be used throughout King's College London (KCL)/King's Health Partners and the research team's social media accounts (e.g., Twitter, Facebook), through internal and external KCL communications and bulletins (e.g., the disability team), and flyers displayed around KCL campuses and other suitable public areas where permission is granted. Flyers and adverts will also be disseminated to the public through charity organisations.

Route 5: Word-of-mouth and snowball sampling. We will invite screened individuals and/or those who have heard about the study to share the study information with their peers.

Randomisation:

Participants will be randomised using King's Clinical Trials Unit's (KCTU) web-based randomisation service. Online peer support requires a sufficiently large community of active users to enable discussion and encourage engagement. We will therefore allocate participants using a 2:1 ratio (100 to the intervention; 50 to control) to maximise the number of participants in the intervention group. Eligible participants will be randomised (T3) following completion of their baseline assessments (T2).

Treatment allocations will be stratified based on depressive symptom severity at baseline using minimisation with randomly varying block sizes. Baseline severity will be measured based on the PHQ-8 total score (Low = PHQ-8 score of <7; High = PHQ-8 score ≥7). Although the research team will be unblind to treatment allocations, the web-based system will conceal subsequent allocations

Intervention:

Through collaboration with people living with LTCs, clinicians, academics, and web design experts, an online peer support and psychoeducation platform to help people with physical health conditions connect, support others, share experiences, and receive evidence-based information and advice on self-management has been co-designed.

The web-based platform offers users access to peer support forums with embedded psychoeducation content. The platform design aims to be inclusive of all people living with LTCs, irrespective of their diagnosis. The inclusive approach that is advocated has been steered by the experiences and vision of our PPI groups. The platform will be moderated throughout the trial.

Control Arm:

Participants in the control arm will be directed towards the "Mental Health" webpage(s), an online resources page provided by the NHS (https://www.nhs.uk/mental-health/). These resources are not specifically targeted at people living with LTCs. They include information sheets and mental health support on topics such as advice for life situations and events. Additionally, it hosts a "self-help" section that includes guides, tools, and activities to support mental health, but does not include any interactive or peer support elements.

Procedures:

The flow of participants through the trial is summarised as follows:

1. Recruitment (T1)
2. Consent to take part in eligibility screenings (T1)
3. First eligibility screening (T1)
4. Wait period
5. Second eligibility screening, consent to trial, baseline assessment (T2)
6. Randomisation (T3)
7. Intervention period (T4)
8. Mid-intervention assessment (T5)
9. Follow-up assessment and qualitative interviews (T6)

After recruitment, individuals will be initially assessed for eligibility via an online questionnaire (T1). Eligible individuals will enter a 'wait period', a delay to allow us to recruit enough participants to open the online platform (i.e., a sufficient number to allow a community to form where discussions can happen). During the wait period, participants can select the frequency of contact they would like to receive from the research team and access a 'live' link summarising recruitment progress. This step was designed following consultations with the RAG. When recruitment targets are met (n=150), all initially eligible individuals (T1) will undergo a second, much shorter, screening assessment (T2) to assess eligibility on time-varying criteria: i) Depressive symptoms (i.e., PHQ-8 score). ii) Diagnosis of bipolar, psychosis, PTSD, and/or schizophrenia or a diagnosis of dementia. We will also invite individuals initially found to be ineligible on time-varying criteria (i) at T1 to be re-screened at T2, since their eligibility may have changed over time. All individuals found to be eligible at the second screening (T2) will be consented, randomised, and invited to complete a baseline assessment (online, via Qualtrics).

Participants will be given two weeks to complete their baseline assessment online. After randomisation, participants in the intervention arm will be invited to join the peer support platform; participants in the control arm will be provided with a link to the NHS "Mental Health" pages. All participants in the intervention arm will be given access to register and create their profile on the platform ahead of the launch date, with all accounts activated on the set "go-live" time (will be determined dependent on recruitment rates). All participants in the control arm will be sent the control condition at the same time as the "go-live" time for the intervention arm. This is to ensure all participants have access to their treatment allocation for the full 3-month period, regardless of when they were randomised. The intervention period will run for three months concurrently for all participants, measured from the date when participant accounts were first activated at the "go-live" timepoint.

Participants will be invited to complete their mid intervention assessment (online via Qualtrics; assessing PHQ-8 and reporting adverse events only) at week six, with a two-week period to complete the questionnaire. After three months, the platform will be closed (no further logins permitted) and participants will be invited to complete a follow-up questionnaire (online via Qualtrics). Participants will be given four weeks (from the end of the intervention period) to return their follow-up questionnaire. In the six weeks after the intervention period, a sample of participants (~30 from intervention arm; ~10 from control arm) will be invited to complete a one-to-one qualitative interview online. All data will be self-reported via online questionnaires (Qualtrics), except for the qualitative interviews. Links to the online questionnaire will be sent to participants via email.

Observational Cohort:

If an individual is ineligible solely due to their PHQ-8 score at T2 (i.e., satisfy the remaining inclusion and exclusion criteria with a PHQ-8 score ≤4 or >9), they will be offered the opportunity to be onboarded onto the peer support platform as part of an observational cohort. We will however exclude those who screen in the ranges of moderate to severe depression (e.g., scores ≥15 on the PHQ-8). These participants will be invited to take part in the community engagement study and have three months of access to the peer support and psychoeducation platform, alongside the participants from the RCT randomised to the intervention arm. All protocols and policies will be the same as those in the intervention arm. This includes a sample of participants being invited to complete qualitative interview at the end of the intervention.

Non-participation:

Patients who initiate contact with the research team (either via consent to contact databases or participant-initiated routes) but subsequently decline to participate in the study will be asked if they would be willing to complete a short anonymous questionnaire about their reasons for non-participation. This will elucidate potential barriers to recruitment and provide data pertaining to the acceptability of the intervention and trial procedures.

Withdrawal:

The intervention is intended to complement the usual care participants receive for their LTCs. Participants can request to withdraw from the intervention at any point, including the closure of their account for those allocated to the peer support platform. In addition, participants may choose to not login (intervention arm) or access the online resources (control arm). The research team will attempt to contact all participants (even those withdrawn from the intervention) to complete follow-up assessments, unless a participant has explicitly requested withdrawal from data collection. There are no criteria for discontinuing or modifying allocated interventions. However, for those participants in the intervention arm, as outlined in the Moderation Policy, access to the platform will be removed under circumstances of severe violations of the Community Principles Users must accept these Community Principles before creating their account on the peer support platform.

Adverse Events:

Adverse events (AEs) and Serious Adverse Events (SAEs) will be captured throughout the three-month trial period. This includes:

1. A self-report questionnaire that will be administered to participants in the intervention arm (CommonGround) and in the control group (NHS Mental Health webpages) at:

   * Six weeks (capturing the initial six weeks of the trial)
   * Three-month follow-up (capturing the second half of the intervention period i.e., weeks 7-12).
2. Monitoring and recording any other SAEs and AEs that occur throughout the three-month trial period as per our study definitions and reporting accordingly.
3. As per recommended guidance on assessing the safety of digital health interventions, monitoring depressive symptom deterioration.

We will work in collaboration with our PPI groups to co-create a list of expected AEs and a text box will be provided to record any other unexpected AEs.

Study End:

This feasibility trial is not powered to assess clinical efficacy, and as such, will not provide conclusions about the potential benefits or safety of the platform. As a result participants will not be permitted to use the platform beyond the three-month intervention period for this reason. End of study will be defined as end of follow-up (i.e. when the last participant has completed their last follow-up/interview).

ELIGIBILITY:
Inclusion Criteria:

* Probable SUBD (scoring 5-9 on the PHQ-8).
* Currently living with one or more LTCs. A long-term condition is a diagnosed physical medical condition with a duration of ≥6 months that demonstrates recurrence or deterioration and is typically associated with a poor prognosis. There are no restrictions on the type of LTCs. Please see list below.
* Aged ≥18 years old.
* Access to the internet (via phone, desktop, or laptop).
* Sufficient English to engage with the platform (assessed via self-report during screening).
* Ability to give informed consent (i.e., no known circumstances/conditions that may affect capacity to consent, e.g., dementia, memory loss or awaiting diagnosis).

Exclusion Criteria:

• Have ever received a clinical diagnosis of severe mental illness of bipolar, psychosis, post-traumatic stress disorder (PTSD), and/or schizophrenia, and/or a diagnosis of dementia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
Incidence of probable Major Depressive Disorder (MDD) | 3 months
  Measured by the Patient Health Questionnaire (PHQ)-8 (PHQ-8 >9 = 1; PHQ-8 ≤9 = 0).

SECONDARY OUTCOMES:
Symptoms of depression | Mid-intervention (Week 6) and 3 months
  Measured by the Patient Health Questionnaire (PHQ)-8 total score. Eight items, each of which is scored 0 to 3, providing a 0 to 24 severity score, with 0 meaning no symptoms and 24 indicating most severe symptoms.
Symptoms of anxiety | 3 months
  Measured by Generalized Anxiety Disorder assessment (GAD-7) total score. Seven items, each of which is scored 0 to 3, providing a 0 to 21 severity score, with 0 meaning no symptoms and 21 indicating most severe symptoms.
Well-being | 3 months
  Measured by the Warwick-Edinburgh Mental Well-Being Scale (WEMWBS). The WEMWBS is scored by summing the scores for each of the 14 items, which are scored from 1 to 5. Minimum score is 5 and maximum is 70, with higher scores indicating greater positive mental wellbeing.
Health-related quality of life | 3 months
  Measured by the Medical Outcomes Study Questionnaire Short Form-36 (SF-36). Scores range from 0-100, with higher scores indicating higher health-related quality of life.
Social connectedness | 3 months
  Measured by the Social Connectedness Scale-Revised (SCS-R). This scale consists of 20 items rated on a scale range from 1 (strongly disagree) to 6 (strongly agree). A higher score indicates more social connectedness to others.
Self-efficacy | 3 months
  Measured by the Chronic Disease Self-Efficacy Scales (CDSES). Each scale is rated from 1-10 with higher numbers indicating higher self-efficacy.
Sense of virtual community | 3 months
  Measured by the Sense of Virtual Community questionnaire (SoVC). Items are rated from 1 = strongly disagree to 7 = strongly agree. Scores are reported as average Likert scales scores with higher scores indicating higher sense of virtual community
Entitativity | 3 months
  An adapted 3-item Entitativity measure. Items are rated from 1 = strongly disagree to 7 = strongly agree. Scores are reported as average Likert scales scores with higher scores indicating higher sense of Entitativity.
Client Services Receipt Inventory (CSRI) | 3 months
  An adapted version of the Client Services Receipt Inventory that measures services and supports that a participant may use over the past 3-month period. Subsections include background demographic information, accommodation and living situation, employment history, health-care service use, and informal supports.
Health Economics | 3 months
  The EQ-5D-5L, a standardised measure of health status, consisting of five dimensions. Standard value sets are summarised using a single index value determining the valuation of health-related quality of life. The numbers representing the five severity levels of a dimension are labels used in the numerical description of a health state. These are not used to determine a summary score. A single index value will be calculated using the preference of the general population in England.

OTHER OUTCOMES:
Feasibility outcomes | Baseline and 3 months
  The primary feasibility outcome will be (1) the number of participants recruited to the trial per week, in total, and for each recruitment route (participants self-report where they heard about the study). Other feasibility outcomes include:
  (2) Number of participants consenting to the eligibility screening(s) of those contacted by the research team via email (e.g., via IMPARTS, Bioresources, Lambeth Talking Therapies; see details below).
  (3) Number of participants found to be eligible at first screening (T1) of those consenting to the eligibility screening(s).
  (4) Number of participants found to be eligible at T2, of those screened at T2. (5) Number of participants giving consent to participate in feasibility trial, of those eligible at T2.
  (6) Number of participants withdrawn from trial, of those randomised. (7) Number of participants responding to follow-up assessment at three months (post-intervention), of those randomised.
Usability | 3 months
  Perceived usability, measured using mHealth App Usability Questionnaire (MAUQ). The MAUQ has demonstrated reliability and validity to measure mHealth App usability. Twenty-one items are presented and rated 1= strongly disagree to 7= strongly agree. The total and average are calculated with the higher the overall average, the higher the usability of the app.
Acceptability | 3 months
  A nested qualitative study will be conducted. Post-intervention qualitative interviews will investigate patients' experiences and views of the peer support platform, including (i) acceptability of the intervention and its perceived benefits and limitations; (ii) acceptability of trial procedures, including views on randomisation, the control condition, and relevance and burden of outcome measures.
Platform adherence - Log-Ins | 3 months
  In the intervention arm only, we will collect data measuring engagement with the peer support platform. This includes clicks and interactions participants make when accessing and using the platform, specifically:
  (1) Number of times logging into the platform (total and per day/week), overall and by device type (e.g., mobile, desktop).
Platform adherence - Duration | 3 months
  In the intervention arm only, we will collect data measuring engagement with the peer support platform. This includes clicks and interactions participants make when accessing and using the platform, specifically:
  (2) Time spent logged in (total and per day/week), overall and by device type (e.g., mobile, desktop).
Platform adherence - Discussion Posts | 3 months
  In the intervention arm only, we will collect data measuring engagement with the peer support platform. This includes clicks and interactions participants make when accessing and using the platform, specifically:
  (3) Number of (i) original posts in the community feed; (ii) comments on posts; (iii) reactions to posts; and (iv) number of searches.
Platform adherence - User Interactions | 3 months
  In the intervention arm only, we will collect data measuring engagement with the peer support platform. This includes clicks and interactions participants make when accessing and using the platform, specifically:
  (4) Number of user-to-user interactions, including (i) follows/unfollows; (ii) 'muting'; (iii) viewing other members' profiles; (iv) number of posts flagged.
Platform adherence - Edited/Deleted Posts | 3 months
  In the intervention arm only, we will collect data measuring engagement with the peer support platform. This includes clicks and interactions participants make when accessing and using the platform, specifically:
  (5) Number of posts edited or deleted by moderators and time spent moderating.
Platform adherence - Content Interactions | 3 months
  In the intervention arm only, we will collect data measuring engagement with the peer support platform. This includes clicks and interactions participants make when accessing and using the platform, specifically:
  (6) Number of times participants (i) download or open resources; and (ii) save content to the 'My Garden' private page.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Hotopf, PhD, FRCPsych, FMedSci, Principal Investigator — King's College London; Elly Aylwin-Foster, MSc, Study Director — King's College London; Ewan Carr, PhD, Study Director — King's College London; Vanessa Lawrence, PhD, Study Director — King's College London; Alan Simpson, PhD, Study Director — King's College London; Ciara Regan, MSc, Study Director — King's College London; Hannah G Jones, BSc, Study Director — King's College London; Grace Lavelle, PhD, Study Director — King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lavelle G, Jones HG, Carr E, Aylwin-Foster E, Lawrence V, Simpson A, Hotopf M. Online Peer Support for Long-Term Conditions: Protocol for a Feasibility Randomized Controlled Trial. JMIR Res Protoc. 2025 Jul 23;14:e71513. doi: 10.2196/71513. PMID 40700748